CLINICAL TRIAL: NCT07404709
Title: Clinical Phase I and IIa Trials of Intratympanic Injection of Small Extracellular Vesicles Derived From Mesenchymal Stem Cells in Severe and Profound Sudden Sensorineural Hearing Loss
Brief Title: Study on the Safety and Efficacy of Intratympanic Injection of Small Extracellular Vesicles Derived From Mesenchymal Stem Cells in Severe and Profound Sudden Sensorineural Hearing Loss
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jiangyan, Chief Physician, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QYFYEC2025-196
Record Dates: First submitted 2025-12-23; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sudden Hearing Loss; Extracellular Vesicles
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group-Clinical Phase I (Experimental): Standard treatment for sudden deafness+hUC-MSC-sEV-003 at low to high dose
  Interventions: Drug: Tympanic injection of hUC-MSC-sEV-003 (small extracellular vesicles) at three different doses
- Control Group--Clinical Phase I (Placebo Comparator): Standard treatment for sudden deafness+hUC-MSC-sEV-003 mimetics
  Interventions: Drug: Standard treatment for sudden deafness+hUC-MSC-sEV-003 mimetics
- Treatment Group--Clinical Phase II (Experimental): Standard treatment for sudden deafness+hUC-MSC-sEV-003 at an appropriate dose as determined by the stage I trial
  Interventions: Drug: Standard treatment for sudden deafness+hUC-MSC-sEV-003 at an appropriate dose as determined by stage I trial
- Control Group--Clinical Phase II (Active Comparator): Standard treatment for sudden deafness+dexamethasone
  Interventions: Drug: Standard treatment for sudden deafness+dexamethasone

INTERVENTIONS:
Drug: Tympanic injection of hUC-MSC-sEV-003 (small extracellular vesicles) at three different doses — In Clinical Phase I, nine participants were additionally injected with small extracellular vesicles at three different doses (low to high concentration，3 participants for each dose) together with traditional drug treatment. The intratympanic injection of small extracellular vesicles was given every other day for a total of 3 times for every participants.
  Arms: Treatment group-Clinical Phase I
Drug: Standard treatment for sudden deafness+hUC-MSC-sEV-003 mimetics — In Clinical Phase I, on the basis of receiving standard treatment for sudden deafness, participants were respectively administered intratympanic injections of hUC-MSC-sEV-003 mimics every other day, with each injection volume being 0.5 ml, for a total of three times.
  Arms: Control Group--Clinical Phase I
Drug: Standard treatment for sudden deafness+hUC-MSC-sEV-003 at an appropriate dose as determined by stage I trial — After the safety verification and dose determination of the Phase I clinical trial were completed, about 20 participants received standard treatment in accordance with the "Guidelines for the Diagnosis and Treatment of Sudden Deafness (2015)", and at the same time, they were administered intratympanic injections of small extracellular vesicles every other day, for a total of 3 times.
  Arms: Treatment Group--Clinical Phase II
Drug: Standard treatment for sudden deafness+dexamethasone — Participants in the control group received standard treatment in accordance with the "Guidelines for the Diagnosis and Treatment of Sudden Deafness (2015)", and during their hospitalization, they received intratympanic injections of dexamethasone at a dose of 5mg every other day for a total of 3 times.
  Arms: Control Group--Clinical Phase II

SUMMARY:
The goal of this clinical trial is to learn if small extracellular vesicles derived from mesenchymal stem cells work to treat severe and above sudden sensorineural hearing loss. It will also learn about the safety of small extracellular vesicles. The main questions it aims to answer are:

1. Does small extracellular vesicles combined with traditional drug treatment improve hearing even better in severe and above sudden deafness participants?
2. What medical problems do participants have with intratympanic injection of small extracellular vesicles? Researchers will compare small extracellular vesicles to dexamethasone to see if small extracellular vesicles work to treat severe and above sudden sensorineural hearing loss.

In clinical Phase I trial, the investigators will complete the safety check and dose exploration.

Participants will:

1. Receive traditional drug treatment in accordance with the "Guidelines for the Diagnosis and Treatment of Sudden Deafness (2015)
2. Receive small extracellular vesicles or a placebo tympanic injection additionally
3. Visit the clinic once every 2 weeks for checkups and tests
4. Receive tympanic injections of small extracellular vesicles ranging from low concentration to high concentration
5. Be evaluated for any adverse reactions In clinical Phase II trial, participants were randomly divided into a control group and an experimental group.

   Participants will:
6. Received intratympanic injections of small extracellular vesicles 3 times together with traditional drug treatment in experimental group
7. Received intratympanic injections of 5mg dexamethasone 3 times together with traditional drug treatment in control group, also for a total of 3 times Visit the clinic once 7 days , 1month and 3 months after treatment for checkups and tests of pure tone audiometry, speech audiometry, tinnitus disability scale and visual analogue scale assessment

ELIGIBILITY:
Inclusion Criteria:

1. Sudden unilateral hearing loss that occurs within 72 hours, with a decrease of at least 30 decibels in at least 3 frequency ranges compared to the healthy ear, and an average pure tone threshold of ≥ 65 decibels.
2. Enrollment must be completed within 7 days after the onset of sudden deafness.
3. Men or women aged 18 to 65
4. Not treated in any other hospital and not taking any treatment medication on one's own
5. Be able to understand the trial protocol and undergo regular follow-up visits and check-ups

Exclusion Criteria:

1. Pregnant or lactating women
2. With a history of chronic ear diseases, ear surgery, autoimmune hearing loss or a confirmed diagnosis of Meniere's syndrome in the past
3. Having received steroid treatment for any reason within the past 30 days
4. There are autoimmune diseases or chronic inflammatory diseases.
5. Severe damage to liver and kidney functions
6. Patients with a previous history of cerebral hemorrhage or those currently taking anticoagulant medications
7. Other cases in which the researchers judged the candidates to be unsuitable for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pure tone test | Baseline,7 days,1 month, and 3 months after clinical phase II treatment
  The hearing recovery status is evaluated based on the changes in pure tone threshold from the baseline at enrollment to 3 months of follow-up. The pure tone threshold is the average of air conduction thresholds at 0.25, 0.5, 1, 2, 4 kHz, and 8 kHz.
speech audiometry | Baseline,7 days,1 month, and 3 months after clinical phase II treatment
  The hearing recovery status is also evaluated based on the changes in speech recognition rate from the baseline at enrollment to 3 months of follow-up. The speech audiometry results use the speech recognition rates at the baseline and after treatment of the subjects.

SECONDARY OUTCOMES:
Respiration | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators monitor vital signs respiration. The unit of respiratory rate is breaths per minute with the normal range 12 to 20 beats per minute.
Heart rate | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators also monitor vital signs heart rate. The unit of heart rate is beats per minute with the normal range 60 to 100 beats per minute at rest.
Oxygen saturation | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators also monitor vital signs oxygen saturation. The unit of oxygen saturation is percent with the normal range of 95% to 100%.
Blood pressure | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators also monitor vital signs blood pressure. The unit of blood pressure is mmHg. The normal range is that the systolic pressure should not exceed 140 mmHg, the diastolic pressure should not exceed 90 mmHg, and the blood pressure level should be no less than 90/60 mmHg.
tympanic membrane healing status | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators observe the healing status of the eardrum. There are two possible outcomes: the eardrum heals or it does not heal.
Haematological index on liver function | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators assess the changes in haematological index on liver function and kidney function levels compared to the baseline. The indicators for evaluating liver function include biochemical indicators such as albumin, transaminases, and bilirubin.
Haematological index on kidney function | Baseline, 2 weeks after intratympanic injection in the first-phase clinical
  The investigators assess the changes in haematological index on kidney function levels compared to the baseline. The indicators for evaluating kidney function include biochemical parameters such as serum creatinine, urea nitrogen, uric acid, glomerular filtration rate, and urine protein.
Tinnitus Handicap Inventory | Baseline,7 days,1 month, and 3 months after clinical phase II treatment
  The assessment of the tinnitus symptoms of the participants is conducted using the Tinnitus Handicap Inventory at both the baseline and different post-treatment periods. This scale classifies tinnitus into four grades as follows: Grade 1 (mild), corresponding to a Tinnitus Handicap Inventory score of 1 to 16. The tinnitus sound is faint and sometimes present, sometimes absent. Grade 2 (moderate), with a Tinnitus Handicap Inventory score of 18 to 36. The tinnitus sound is relatively obvious but generally has a minor impact. Grade 3 (moderately severe), with a Tinnitus Handicap Inventory score of 38 to 56. The tinnitus sound is moderate and begins to cause some interference in daily life. Grade 4 (severe), with a Tinnitus Handicap Inventory score of 58 to 76. A higher score means a worse result.
Visual Analogue Scale | Baseline,7 days,1 month, and 3 months after clinical phase II treatment
  The psychological assessment of the participants is carried out using the Visual Analogue Scale.The VAS scoring standard uses a straight line or ruler approximately 10 centimeters long, with the two ends marked as 0 and 10 respectively. 0 indicates no pain, and 10 indicates severe pain. Participants mark the corresponding position according to the degree of pain. 2. Pain grading: 0 indicates no pain; 1-3 indicates mild pain; 4-6 indicates moderate pain; 7-9 indicates severe pain; 10 indicates extreme pain. In this scale，a higher score means a worse result.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - he Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Chongqing General Hospital, Chongqing, Sichuan

IPD SHARING:
Plan to Share IPD: No
The informed consent form of this study does not include clauses authorizing IPD sharing. As a Phase I/II exploratory study, the data involves sensitive medical information and preliminary research results. To protect participants' privacy and comply with ethical and regulatory requirements, the data will not be shared.